CLINICAL TRIAL: NCT01438710
Title: Switching Study of Kidney Transplant Patients With Tremor to LCP-Tacro (STRATO)
Acronym: STRATO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCP-Tacro 3003
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Renal Failure; Tremors
MeSH Terms: conditions — Renal Insufficiency; Tremor | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCP-Tacro (Experimental): LCP Tacro tables for once daily oral administration
  Interventions: Drug: LCP-Tacro
- Prograf (Experimental): Tacrolimus capsules for twice daily oral administration
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Prograf — Oral Prograf or generic tacrolimus doses will be taken b,i,d, consistently in 2 divided doses, once in the morning and once in the evening, to maintain trough level in the range of 3 to 12 ng/mL. Target trough level for the subject will be determined per clinical practice.
  Other Names: tacrolimus
  Arms: Prograf
Drug: LCP-Tacro — LCP-Tacro will be administered orally q.d. in the morning based on a conversion factor from Prograf or generic tacrolimus to LCP-Tacro of 0.7 for non-African American subjects and 0.85 for African American subjects to maintain target trough level of 3 to 12 ng/mL.
  Other Names: tacrolimus
  Arms: LCP-Tacro

SUMMARY:
This study will evaluate and measure symptomatic hand tremor in stable kidney transplant subjects on Prograf or generic tacrolimus maintenance therapy at baseline (pre-conversion) and following conversion to LCP-Tacro. This study will also evaluate the safety of LCP-Tacro compared with Prograf or generic tacrolimus

DETAILED DESCRIPTION:
This is a 2 sequence, open-label, multicenter, prospective Phase 3b clinical study to access drug-induced hand tremors in stable kidney transplant subjects converted from Prograf (tacro-limus, Astellas Pharma US, Inc., Deerfield, IL) or generic tacrolimus twice daily (b.i.d.) to LCP-Tacro tablets (tacrolimus, Veloxis Pharmaceuticals A/S, Horsholm, Denmark) once daily (q.d.). The trial is designed to determine if the test drug LCP-Tacro, is associated with fewer and/or less severe drug-induced hand tremor than observed with Prograf or generic tacrolimus treatment; each therapy is to be concomitantly administered with mycophenolate mofetil (MMF), mycophenolate sodium (MPS), including generic versions of each, and/or prednisone or equivalent as long as doses remain stable during the study. All prophylaxis and other medication will be allowed per standard of care (SOC) in each of the participating sites; no medication that interacts with the pharmacokinetics (PK) of tacrolimus is allowed unless subjects who are recipients of a renal transplant at least 1 month and not more than 5 years prior to enrollment. Following screening, study visits will be conducted over a 2-week treatment period with consists of 1 week of Prograf or generic tacrolimus SOC, and 1 week of LCP-Tacro. Subjects who qualify for extended use of LCP-Tacro can continue LCP-Tacro treatment for additional 2 years. This decision will be made at the discretion of the physician and subject.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to give written consent
2. Men and women between 18 and 65 years of age who are recipients of a kidney transplant between 1 month and 5 years prior to the screening date
3. Subjects with at least one complaint of tremor and existence of postural tremor or action tremor on finger to nose as demonstrated by a score of at least 2 of any of the 4 upper extremity (UE) postural or action and intention assessments on the FTM clinical rating scale
4. Subjects experiencing symptomatic drug-induced hand tremor associated with use of Prograf or generic tacrolimus as demonstrated by responding "no" to each of the following question: "Did you have a tremor that you noticed prior to starting Prograf or generic tacrolimus for your kidney transplant?", or "Are you aware of a tremor that runs in your family?"
5. Subjects taking a stable dose of oral Prograf or generic tacrolimus capsules for at least 7 days with trough levels of tacrolimus between 3 to 12 ng/mL. Subjects must maintain tacrolimus trough levels in this range during the 7 day Prograf or generic tacrolimus treatment phase (note that 1 dose adjustment at Study Day 3 [a.m.dose] is allowed for those subjects whose Day0/1 trough level is out of range.
6. Women of childbearing potential must have a negative serum pregnancy test within 7 days before study start.

Exclusion Criteria:

1. Recipients of any transplants including organ other than kidney and bone marrow
2. Subjects with an estimated glomerular filtration rate (eGFR) (MDRD7) <30mL/min at Screening
3. Subjects incapable of understanding the purposed and risks of the study, who cannot give written informed consent and who are unwilling or unable to comply with study protocol requirements
4. Pregnant or nursing women
5. Subjects with reproductive potential who are unwilling/unable to use a double barrier method of contraception
6. Subjects who were treated with any other investigational agent within 3 months prior to screening
7. Subjects who are taking drugs that are likely to affect the PK levels of tacrolimus and are not on a stable dose of those medications (see Appendix 1)
8. Subjects who have essential tremor, Parkinsonism, or tremor from any cause other than tacrolimus-induced tremor;
9. Subjects who are taking or had been taking any drug within the past 30 days that is well known to promote tremors, including: amiodarone, beta-agonist inhalers (such as albuterol), cyclosporine, lithium, metoclopramide, theophylline, or valproate,or taking within the past 6 months the dopamine blocking agents (antipsychotics) (note, other such medication may be considered on a case-by-case basis at the discretion of the investigator);
10. Subjects who taking drugs that reduce tremor, and are not on stable doses of the treatment (ie, had not been taking the medication for a minimum of 30 days), including: gabapentin (note, other such medications may be considered on a case-by-case basis at the discretion of the investigator);
11. Subjects on concurrent immunosuppression with MMD (CellCept) of MPS delayed-release tables (Myfortic), or generic versions of these medication, who have not been on stable doses at least 7 days prior to screening
12. Subjects receiving prednisone or equivalent at a dose >10 mg per day
13. Either subjects with an episode of acute rejection requiring treatment or subjects with an episode of biopsy-proven or suspected acute rejections that requires treatment within 3 months of screening
14. Subjects who are being actively treated for cancer (with the exception of non-invasive basal cell or squamous cell) or human immunodeficiency virus (HIV)
15. Subjects with any form of current drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Glicklich, MD, Study Director — VP, Clinical Development
Locations (10):
- United States (10):
  - Clinical Investigative Site 006, Los Angeles, California
  - Clinical Investigative Site 1049, San Diego, California
  - Clinical Investigative Site 007, Aurora, Colorado
  - Clinical Investigative Site 005, New Haven, Connecticut
  - Clinical Investigative Site 004, Lexington, Kentucky
  - Clinical Investigative Site 008, Minneapolis, Minnesota
  - Clinical Investigative Site 003, St Louis, Missouri
  - Clinical Investigative Site 002, Oklahoma City, Oklahoma
  - Clinical Investigative Site 009, Nashiville, Tennessee
  - Clinical Investigative Site 012, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- LCP-Tacro: After the first weeks treatment with Prograf/generic Tacrolimus, all patients were switched to LCP Tacro tables for once daily oral administration for one week.
  LCP-Tacro: LCP-Tacro will be administered orally q.d. in the morning based on a conversion factor from Prograf or generic tacrolimus to LCP-Tacro of 0.7 for non-African American subjects and 0.85 for African American subjects to maintain target trough level of 3 to 12 ng/mL.
- Prograf: All patients received Prograf/generic Tacrolimus capsules for twice daily oral administration during the first week of treatment.
  Prograf: Oral Prograf or generic tacrolimus doses will be taken b,i,d, consistently in 2 divided doses, once in the morning and once in the evening, to maintain trough level in the range of 3 to 12 ng/mL. Target trough level for the subject will be determined per clinical practice.
Period: First Week of Treatment
Arm/Group | LCP-Tacro | Prograf
Started | 0 (Patients are only treated with Prograf/generic Tacrolimus during the first week.) | 44
Completed | 0 (Patients are only treated with Prograf/generic Tacrolimus during the first week.) | 41
Not Completed | 0 | 3
Period: Second Week of Treatment
Arm/Group | LCP-Tacro | Prograf
Started | 41 (Patients completing the first week will continue on LCP-Tacro treatment during the second week.) | 0 (Patients are only treated with LCP-Tacro during the second week.)
Completed | 40 | 0 (Patients are only treated with LCP-Tacro during the second week.)
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: 44 patients started on the initial one-week treatment on Prograf and 41 were switched to the one-week LCP-Tacro treatment. 40 patients completed the one-week treatment on LCP-Tacro and continued into the 24-months extended use period.
Arm/Group | Prograf
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 34
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 44
Target Trough Range (low), ng/mL [Mean (Standard Deviation); unit: ng/mL] | 5.72 (1.912)
Target Trough Range (high), ng/mL [Mean (Standard Deviation); unit: ng/mL] | 8.68 (1.863)
Height, cm [Mean (Standard Deviation); unit: cm] | 173.63 (8.424)
Weight, kg [Mean (Standard Deviation); unit: kg] | 88.16 (19.707)
BMI, kg/m2 [Mean (Standard Deviation); unit: kg/m2] | 29.20 (5.979)
Time from current kidney transplant to enrolment, months [Mean (Standard Deviation); unit: Months] | 16.85 (14.455)
Donor type for current kidney transplant, n [Number; unit: participants]
  Living donor | 15
  Deceased donor | 29

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Hand Tremor and Stable Kidney Transplant Patients When Switched From Prograf to LCP-Tacro.
Description: The primary efficacy endpoint is the mean change from baseline (ie Day 7) in the Fahn-Tolosa-Marin Clinical Rating Scale (FTM) for overall tremor score 7 days after (ie, Day 14) LCP-Tacro conversion.
  The overall FTM score was 0 to 100 where higher scores denoted worst/more severe tremor.
  Below the mean total score and standard deviation for each treatment is given in addition to the mean change.
Time Frame: 14 days
Population: Of the 40 patients who completed the study period, 38 patients were evaluable for efficacy evaluation and included in the modified intention to treat (mITT) population.
  The outcome measure is given as total score below.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 38
units on a scale
  Total score day 7 (Prograf) | 25.30 (9.472)
  Total score day 14 (LCP-Tacro) | 19.96 (7.613)
  Mean change | -5.35 (7.501)
Statistical Analysis 1: Comparison: LCP-Tacro; The mean change (i.e., absolute change) from baseline (Day 7, pre-conversion) on FTM overall score to Day 14 (post-conversion) was evaluated using paired t-test (at 0.05 significance level, two sided). An estimation of mean change from baseline and the corresponding 95% confidence interval (CI) were provided; Test type: Superiority or Other; p = 0.0048, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Each patient was followed for 25 months.
Description: AE threshold is defined as 5% per treatment arm; i.e. at least 2 patients in the treatment arm have experienced the event.
Arm/Group | LCP-Tacro | Prograf
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/44
Other Adverse Events (participants affected / at risk) | 2/41 | 7/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=41) | Prograf (N=44)
Incision Site Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=41) | Prograf (N=44)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Cardiac Murmur (Investigations) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other